CLINICAL TRIAL: NCT05093972
Title: An Open-Label, Single-Dose Clinical Study to Evaluate Pharmacokinetics of MK-8507 in Participants With Mild or Moderate Hepatic Impairment.
Brief Title: Ulonivirine (MK-8507) in Participants With Mild or Moderate Hepatic Impairment (MK-8507-014)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8507-014; MK-8507-014 (Other: MSD)
Record Dates: First submitted 2021-10-18; First posted 2021-10-26 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — ulonivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Panel A: Mild HI (Experimental): Participants with mild HI receive a single oral dose of ulonivirine 400 mg on Day 1.
  Interventions: Drug: Ulonivirine
- Panel B: Moderate HI (Experimental): Participants with moderate HI receive a single oral dose of ulonivirine 400 mg on Day 1.
  Interventions: Drug: Ulonivirine
- Panel C: Healthy Controls (Active Comparator): Healthy matched control participants receive a single oral dose of ulonivirine 400 mg on Day 1.
  Interventions: Drug: Ulonivirine

INTERVENTIONS:
Drug: Ulonivirine — Four ulonivirine 100 mg tablets (total dose 400 mg) taken by mouth.
  Other Names: MK-8507

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics (PK) and safety of a single oral dose of ulonivirine in participants with mild or moderate hepatic impairment (HI). It is hypothesized that the area under the plasma concentration-time curve from dosing to (extrapolated) infinity (AUC0-∞) in participants with mild or moderate HI is similar to that of healthy control participants.

ELIGIBILITY:
Inclusion Criteria:

Mild and Moderate HI (Panels A and B):

* Has a diagnosis of chronic (>6 months), stable HI with features of cirrhosis due to any etiology (stability of hepatic disease should correspond to no acute episodes of illness within the previous 2 months due to deterioration in hepatic function)

Healthy Controls (Panel C):

* Is in good health

All Participants (Panels A to C):

* Has a body mass index (BMI) ≥18.5 and ≤40 kg/m^2, inclusive
* If male, uses contraception in accordance with local regulations
* If female, is not pregnant or breastfeeding and one of the following applies: 1) is not a woman of childbearing potential (WOCBP), or 2) is a WOCBP and is abstinent/uses acceptable contraception, has a negative highly sensitive pregnancy test within 24 hours of receiving study intervention, and provides medical/menstrual/recent sexual history for review by the investigator

Exclusion Criteria:

Mild and Moderate HI (Panels A and B):

* Has a history of any illness that, in the opinion of the investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study
* Is not in sufficient health
* Is institutionalized/mentally or legally incapacitated
* Is positive for human immunodeficiency virus (HIV)-1 or HIV-2
* Has received antiviral and/or immune modulating therapy for hepatitis B virus (HBV) or hepatitis C virus (HCV) within 90 days prior to study start
* Is taking medication for a chronic condition and has not been on a stable regimen for ≥ 1 month

Healthy Controls (Panel C):

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated
* Is positive for hepatitis B virus surface antigen (HBsAg), hepatitis C antibodies, HIV-1, or HIV-2
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to first dose of study drug

All Participants (Panel A to C):

* Has a history of cancer (malignancy)
* Has a history of significant multiple and/or severe allergies
* Has known hypersensitivity to the active substance or any of the excipients of the study drug
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-04-07 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Dosing to Infinity (AUC0-∞) of Ulonivirine | Predose and 1, 2, 4, 6, 8, 12, 24, 48, 96, 120, 168, 240, 336, and 504 hours postdose
  The AUC0-∞ of ulonivirine will be determined in participants with mild or moderate HI and healthy controls.
Area Under the Plasma Concentration-Time Curve from Dosing to Last Measurable Concentration (AUC0-last) of Ulonivirine | Predose and 1, 2, 4, 6, 8, 12, 24, 48, 96, 120, 168, 240, 336, and 504 hours postdose
  The AUC0-last of ulonivirine will be determined in participants with mild or moderate HI and healthy controls.
Maximum Plasma Concentration (Cmax) of Ulonivirine | Predose and 1, 2, 4, 6, 8, 12, 24, 48, 96, 120, 168, 240, 336, and 504 hours postdose
  The Cmax of ulonivirine will be determined in participants with mild or moderate HI and healthy controls.
Time to Maximum Plasma Concentration (Tmax) of Ulonivirine | Predose and 1, 2, 4, 6, 8, 12, 24, 48, 96, 120, 168, 240, 336, and 504 hours postdose
  The Tmax of ulonivirine will be determined in participants with mild or moderate HI and healthy controls.
Apparent Plasma Terminal Half-life (t½) of Ulonivirine | Predose and 1, 2, 4, 6, 8, 12, 24, 48, 96, 120, 168, 240, 336, and 504 hours postdose
  The t½ of ulonivirine will be determined in participants with mild or moderate HI and healthy controls.
Apparent Total Clearance from Plasma After Oral Administration (CL/F) of Ulonivirine | Predose and 1, 2, 4, 6, 8, 12, 24, 48, 96, 120, 168, 240, 336, and 504 hours postdose
  The CL/F of ulonivirine will be determined in participants with mild or moderate HI and healthy controls.
Apparent Volume of Distribution during Terminal Phase (Vz/F) of Ulonivirine | Predose and 1, 2, 4, 6, 8, 12, 24, 48, 96, 120, 168, 240, 336, and 504 hours postdose
  The Vz/F of ulonivirine will be determined in participants with mild or moderate HI and healthy controls.

SECONDARY OUTCOMES:
Percentage of Participants with an Adverse Event (AE) | Up to 21 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/